CLINICAL TRIAL: NCT00581412
Title: Composite Graft Use in Abdominal Sacrocolpopexy Reduces Erosion Rates
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Karen Noblett, Associate Professor, University of California, Irvine Medical Center
Other Study IDs: 2007-5858
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Composite biologic/synthetic graft; Abdominal sacrocolpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to determine whether the use of a composite biologic/synthetic graft during abdominal sacrocolpopexy leads to a lower rate of erosion while maintaining durability.

DETAILED DESCRIPTION:
This study will examine the erosion rate of a composite graft that is being used during abdominal sacrocolpopexy. The composite graft is composed of a dual layer of biological and syntheric material. Biological grafts have the advantage of significantly reducing erosion rates, but the longevity of biologic graft is uncertain. On the other hand, synthetic grafts have the advantage in that they are durable, but have higher erosion rates through the vagina and require re-operation in a small percentage of patients. This study will look at whether or not the use of a composite greaft carries the advantages of both types of materials and leads to decreased rates of erosion while maintaining longevity. The cost effectiveness of this new type of graft will also be reviewed since the disavantage of utilizing both the synthetic and biologic graft is that it will increase the cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent abdominal sacrocolpopexy with Drs. Noblett and Lane from 2001 to present

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent abdominal sacrocolpopexy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The erosion rates of composite biologic/syntheric grafts and synthetic-only grafts will be compared. | To the point of graft erosion after abdominal sacrocolpopexy

SECONDARY OUTCOMES:
Cost effectiveness will be examined by comparing the price of a composite graft to the cost of re-operation due to erosion of a synthetic-only graft. | To the point of graft erosion after abdominal sacrocolpopexy

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States